CLINICAL TRIAL: NCT07351019
Title: Colonoscopy Bowel Prep Comparison Among Diabetic Patients: Golytely v. SUPREP
Brief Title: Colonoscopy Bowel Prep Comparison Among Diabetic Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eisenhower Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Darrell F. Barker, MD, FACG, Principal Investigator, Eisenhower Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: DDEAMC.2022.0044
Record Dates: First submitted 2026-01-15; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Colon Cancer Screening
MeSH Terms: interventions — Golytely

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Diabetic patients undergoing bowel prep for screening colonoscopy using Golytely (Active Comparator)
  Interventions: Drug: Golytely
- Diabetic patients undergoing bowel prep for screening colonoscopy using SUPREP (Active Comparator)
  Interventions: Drug: SUPRPEP

INTERVENTIONS:
Drug: Golytely — Bowel cleanliness and patient tolerability
  Arms: Diabetic patients undergoing bowel prep for screening colonoscopy using Golytely
Drug: SUPRPEP — Bowel cleanliness and patient tolerability
  Arms: Diabetic patients undergoing bowel prep for screening colonoscopy using SUPREP

SUMMARY:
The goal of this clinical trial is to learn if the Golytely or SUPREP bowel preparation works more effectively in bowel cleansing for colorectal cancer screening with colonoscopy in patients with diabetes. The main questions this study aims to answer are:

1. Is there a significant difference in bowel prep cleanse between Golytely and SUPREP in patients with diabetes based on the Boston Bowel Prep Score (BBPS) as assessed by blinded, skilled endoscopists?
2. Is there a significant difference in patients' tolerance between the bowel preparations as assessed by the validated Mayo Bowel Prep Tolerability Form (MBPTF)?

Participants will:

* Be randomized to take either Golytely or SUPREP bowel preparation prior to their colonoscopy
* Complete the MBPTF on the procedure date prior to the scheduled colonoscopy
* Undergo a standardized screening colonoscopy during which time a blinded endoscopist will document the participant's BBPS

The research team hypothesizes that SUPREP will have a significant difference in tolerability (based on MBPTF), while exhibiting no difference in bowel cleanse (based on BBPS) in the diabetic patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Participants having provided informed consent with signature on informed consent form: the informed consent process should be complete with full discussion of all requirements and possible risks.
2. Diabetic volunteer (defined per current ACP guidelines, and any type of DM)
3. Aged 18+ years, inclusive
4. Average screening risk, polyp surveillance, and family history of cancer

Exclusion Criteria:

1. Unable to provide informed consent to participate in the study Such as a mental condition rendering the participant unable to understand the nature, scope, and possible consequences of the study
2. Clinically relevant cardiovascular, hepatic, neurological, endocrine, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult or that would put the participant at risk by participating in the study
3. Persistent significant or severe infection, either acute or chronic
4. Prior use of any investigational drug in the preceding 6 months
5. Liver function impairment or persisting elevations (confirmed by retest) of alanine aminotransferase (ALT), aspartate aminotransferase (AST), or direct bilirubin greater than 2x the upper limit of normal range (ULN).
6. Pregnant or breast-feeding women or those who plan to become pregnant during the study
7. Participants with significantly impaired bone marrow function or significant anemia, leukopenia, or thrombocytopenia (confirmed by retest):

   1. Hematocrit < 35% and/or
   2. Absolute white blood cell count < 3000 cells/mm3 ( L) and/or
   3. Platelet count < 150 000 cells/mm3 ( L) and/or- Absolute neutrophil = 1500 cells/mm3 ( L)
8. History of colorectal cancer
9. Inflammatory Bowel Disease
10. Past surgical history of colon resection
11. Prior history of colorectal surgery
12. Family history of hereditary polyposis and cancer disorders to include but not limited to FAP (Familial Adenomatous Polyposis), Gardner Syndrome, Turcot Syndrome, Lynch Syndrome, Cowden Syndrome, and Peutz-Jeghers Syndrome
13. Symptomatic patients (bleeding, diarrhea, constipation, abdominal pain)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-16 (Estimated); Primary Completion 2026-07-28 (Estimated); Study Completion 2026-07-28 (Estimated)

PRIMARY OUTCOMES:
Bowel cleanliness using the Boston Bowel Prep Score (BBPS) | Procedural (during the participant's screening colonoscopy)
  The BBPS uses a score from 0-9 which helps quantify bowel cleanliness after bowel prep prior to colonoscopy. A higher score indicates better visualization of the colon mucosa. This will be assessed by blinded, skilled endoscopists.
Use of the Mayo Bowel Prep Tolerability Score (MTS) | Pre-procedural (prior to the participant's screening colonoscopy)
  The questionnaire is a validated scoring system used to assess the tolerability (ex. symptoms) and experience (ex. likelihood of using the bowel prep again) among diabetic patients undergoing the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Dwight D. Eisenhower Army Medical Center, Fort Gordon, Georgia, United States